CLINICAL TRIAL: NCT03468725
Title: A Double-blind, Placebo-controlled Crossover Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Effects on Transcranial Magnetic Stimulation of Oral Administration of XEN1101 in Healthy Male Subjects
Brief Title: Safety, Tolerability, Pharmacokinetics and Effects on Transcranial Magnetic Stimulation of Oral Doses of XEN1101
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xenon Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: XPF-008-101b; 2017-003181-27 (EudraCT Number); C17047 (Other: Richmond Pharmacology's Study Code)
Record Dates: First submitted 2018-03-02; First posted 2018-03-16 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Healthy Male Volunteers
Keywords: Transcranial magnetic stimulation
MeSH Terms: interventions — microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XPF-008 (Experimental): Single oral dose
  Interventions: Drug: XPF-008
- Placebo (Active Comparator): Single oral dose
  Interventions: Drug: Microcrystalline Cellulose

INTERVENTIONS:
Drug: XPF-008 — Capsule filled with XEN1101
  Arms: XPF-008
Drug: Microcrystalline Cellulose — Placebo capsule
  Arms: Placebo

SUMMARY:
The XEN1101 Phase 1 clinical trial is a randomized, double-blind, placebo-controlled study that will eventuate the safety, tolerability, pharmacokinetics (PK) and effects on transcranial magnetic stimulation (TMS) of oral doses of XEN1101 in healthy male subjects.The TMS procedure is designed to demonstrate delivery of XEN1101 into the central nervous system and to observe a change in cortical excitability as measured by EEG and/or EMG activity. It is estimated there will be approximately 15 subjects in the planned study.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy male aged between 18 and 55 years inclusive with a body mass index (BMI) between 18.5 and 30.0 kg/m2
* Right-handed only
* Must agree to use effective methods of contraception, if applicable
* Able to swallow multiple capsules
* Able to provide written, personally signed and dated Informed Consent Form

Key Exclusion Criteria:

* Any current and relevant history of significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk, affect clinical or laboratory results, or the subject's ability to participate in the study
* Any clinically significant abnormalities in vital signs, ECGs, physical examinations, or laboratory evaluations
* Answering "yes" to any of the questions within the Columbia Suicide Severity Rating Scale Mental incapacity or language barriers precluding adequate understanding, cooperation, and compliance with the study
* No prescription or over-the-counter (OTC) medications (including multivitamins, herbal or homeopathic preparations 14 days or if applicable/available, 5 half-lives prior to dosing to study end
* Any history of severe head trauma
* No smoking 60 days prior to dosing to study end

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-02-13 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) as assessed by CTCAE v4.03 | From screening (28 days prior to Day 1) through to 30 days post-final dose
  To assess AEs as a criteria of safety and tolerability
Resting 12-lead electrocardiogram (ECG) | From screening (28 days prior to Day 1) through to Day 14
  To assess ECG intervals (PR, QRS, QTcF, RR) as a criteria of safety and tolerability
Number of participants with vital sign abnormalities | From screening (28 days prior to Day 1) through to Day 14
  To assess vital signs as a criteria of safety and tolerability
Pharmacodynamic (PD) Effects assessed by Transcranial Magnetic Stimulation (TMS) biological markers of brain excitability | Day 1 predose through to Day 7
  To assess biological marker of brain excitability: amplitude (in uV) of TMS evoked potentials on the EEG
PD Effects assessed by TMS biological markers of brain excitability | Day 1 predose through to Day 7
  To assess biological marker of brain excitability: resting motor threshold (in %) for elicitation of an electromyographic response

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Day 1 predose through to Day 8
  Cmax is the maximum observed plasma concentration in ng/mL
Terminal elimination half-life (t1/2) | Day 1 predose through to Day 8
  The time in hours required for the plasma level of the study drug to decrease by one-half during the terminal elimination phase
Area Under the Plasma Concentration-Time Curve from Time Zero to the Time of the Last Quantifiable Plasma Concentration (AUC0-last) | Day 1 predose through to Day 8
  The area under the plasma concentration-time curve [in ng.h/mL] from time zero to the time corresponding to the last quantifiable plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Beatch, PhD, Study Director — Xenon Pharmaceuticals Inc.
Locations (1):
- King's College Hospital, Brixton, London, United Kingdom